CLINICAL TRIAL: NCT04502654
Title: Postoperative Functional Recovery After Fast-track VATS Lobectomy
Brief Title: Rehabilitation for Thoracoscopic Lobectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lin Huang, Medical Doctor, Research fellow, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-20041489
Record Dates: First submitted 2020-07-31; First posted 2020-08-06 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms; Rehabilitation; Exercise; Pain, Postoperative; Post Discharge
Keywords: Functional recovery; Enhanced recovery after surgery; Video-assisted thoracoscopic surgery; Lobectomy
MeSH Terms: conditions — Lung Neoplasms; Motor Activity; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pilot group: As a pilot Group for observating variable rehabilitation under individual baselines.
  Interventions: Device: Actiwatch 2 (Philips Respironics, Murrysville, USA)

INTERVENTIONS:
Device: Actiwatch 2 (Philips Respironics, Murrysville, USA) — Actiwatch 2 is an unobtrusive, waterproof, light sensor and wrist-worn device (weight 16.0g, size 4.3 cm* 2.3 cm* 1.0 cm), containing a tri-axial accelerometer able to records a digitally integrated measure of gross motor activity (a piezoelectric sensor to detect vertical accelerations at the wrist between 0.5 and 2.0 g with a frequency response range between 0.35-7.5 Hz). Activity counts from the device reflect the peak acceleration detected over each epoch and are used in determining sleep and wake intervals, which can be used to rest-activity patterns, quality of physical activity and sleep for 15-60 seconds/ epoch, 24 hours/ day, 2 weeks.

SUMMARY:
The main aim of this research is to compare the functional recovery after discharge with the preoperative physical activity as a hypothesis generating study.

ELIGIBILITY:
Inclusion Criteria:

* VATS-L
* Speaks and understands Danish or English.
* Informed consent obtained

Exclusion Criteria:

* Co-VATS-L.
* on the wheelchair.
* Living in nurse home.
* Using rollator to assist to walk.
* Unwilling to place the Actiwatch 2 or execute PPE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be submitted to video-assisted thoracoscopic surgery lobectomy.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Length of functional rehabilitation | Through study completion, minimum 7 days
  Investigators will calculate preperative Activity Counts per day as a baseline then being compared to postoperative Activity Counts per day until one day when both Counts is equal. Length of functional rehabilitation defines that duration from surgical day to the day when both Counts is equal.

SECONDARY OUTCOMES:
Quality of recovery | Through study completion, an average of 14 days
  The translation of the Danish version of the postoperative quality of recovery scale QoR-15D is used to evaluate the quality of care.
The quantization of fatigue | Through study completion, an average of 14 days
  The Christensen Fatigue Scale (ChrFS) will be utilized to evaluate the degree of fatigue.
The quantization of pain | Through study completion, an average of 14 days
  The numeric rating scale (NRS) ranging from 0 (no pain) to 10 (excruciating pain) is used to score postoperative pain.
The quantization of vomiting. | Through study completion, an average of 14 days
  The numeric rating scale (NRS) ranging from 0 (nothing) to 10 (worest) is used to score postoperative vomiting.
The quantization of nausea. | Through study completion, an average of 14 days
  The numeric rating scale (NRS) ranging from 0 (nothing) to 10 (worest) is used to score postoperative nausea.
The quantization of Activity Counts | Through study completion, an average of 14 days
  Investigators will use Electric Devices to record Activity Counts per day. Activity counts will be classified as sedentary behavior (SB) < 1303 counts/min (cpm), low intensity physical activity (LIPA) 1303 cpm - < 2588 cpm, and moderate to vigorous physical activity (MVPA) ≧2588 cpm.
Length of sleep time | Through study completion, an average of 14 days
  Investigators will use devices to record the specific sleep time for patients.
The quantization of morbidity | up to 30 days
  The Clavien-Dindo Classification (CDC) is applied as a standard to grade the morbidity in 30 days after surgery.
The quantization of mortality | up to 30 days
  Investigators will investigate whether patients will experience unexpected death in 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lin Huang, MD, Principal Investigator — Rigshospitalet, Denmark; Henrik Kehlet, Professor, MD, DMSc, Study Director — Rigshospitalet, Denmark; Rene H Petersen, Professor, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Background] Yang CJ, Kumar A, Deng JZ, Raman V, Lui NS, D'Amico TA, Berry MF. A National Analysis of Short-term Outcomes and Long-term Survival Following Thoracoscopic Versus Open Lobectomy for Clinical Stage II Non-Small-Cell Lung Cancer. Ann Surg. 2021 Mar 1;273(3):595-605. doi: 10.1097/SLA.0000000000003231. PMID 30946089
- [Background] Marijic P, Walter J, Schneider C, Schwarzkopf L. Cost and survival of video-assisted thoracoscopic lobectomy versus open lobectomy in lung cancer patients: a propensity score-matched study. Eur J Cardiothorac Surg. 2020 Jan 1;57(1):92-99. doi: 10.1093/ejcts/ezz157. PMID 31157367
- [Background] Iwata H, Shirahashi K, Yamamoto H, Marui T, Matsumoto S, Mizuno Y, Matsumoto M, Mitta S, Miyamoto Y, Komuro H. Propensity score-matching analysis of hybrid video-assisted thoracoscopic surgery and thoracoscopic lobectomy for clinical stage I lung cancerdagger. Eur J Cardiothorac Surg. 2016 Apr;49(4):1063-7. doi: 10.1093/ejcts/ezv296. Epub 2015 Aug 30. PMID 26324682
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Kehlet H. Enhanced postoperative recovery: good from afar, but far from good? Anaesthesia. 2020 Jan;75 Suppl 1:e54-e61. doi: 10.1111/anae.14860. PMID 31903577
- [Background] Wang KY, Chang NW, Wu TH, Hsu CC, Lee YH, Lee SC. Post-discharge health care needs of patients after lung cancer resection. J Clin Nurs. 2010 Sep;19(17-18):2471-80. doi: 10.1111/j.1365-2702.2010.03298.x. PMID 20920075
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Factors determining convalescence after uncomplicated laparoscopic cholecystectomy. Arch Surg. 2001 Aug;136(8):917-21. doi: 10.1001/archsurg.136.8.917. PMID 11485527
- [Background] Luna IE, Kehlet H, Wede HR, Hoevsgaard SJ, Aasvang EK. Objectively measured early physical activity after total hip or knee arthroplasty. J Clin Monit Comput. 2019 Jun;33(3):509-522. doi: 10.1007/s10877-018-0185-5. Epub 2018 Jul 23. PMID 30039461
- [Background] Aasvang EK, Luna IE, Kehlet H. Challenges in postdischarge function and recovery: the case of fast-track hip and knee arthroplasty. Br J Anaesth. 2015 Dec;115(6):861-6. doi: 10.1093/bja/aev257. Epub 2015 Jul 25. PMID 26209853
- [Background] Timmerman JGJ, Dekker-van Weering MGHM, Wouters MWJMM, Stuiver MMM, de Kanter WW, Vollenbroek-Hutten MMRM. Physical behavior and associations with health outcomes in operable NSCLC patients: A prospective study. Lung Cancer. 2018 May;119:91-98. doi: 10.1016/j.lungcan.2018.03.006. Epub 2018 Mar 9. PMID 29656759
- [Background] Wolvers MDJ, Bussmann JBJ, Bruggeman-Everts FZ, Boerema ST, van de Schoot R, Vollenbroek-Hutten MMR. Physical Behavior Profiles in Chronic Cancer-Related Fatigue. Int J Behav Med. 2018 Feb;25(1):30-37. doi: 10.1007/s12529-017-9670-3. PMID 28699090